CLINICAL TRIAL: NCT06129838
Title: Investigation of Inflammation in Alzheimer's Disease and Related Dementias (ADRD) Using [11C]-CS1P1
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology Division, Diagnostic Radiology Section, Neuroradiology, Washington University School of Medicine
Other Study IDs: CS1P1-ADRD
Record Dates: First submitted 2023-11-01; First posted 2023-11-13 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — sphingosine 1-phosphate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for future research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Healthy participants will receive a single intravenous bolus injection of 12.0 - 17.0 milliCurie (mCi) of the investigational radiotracer [11C]-CS1P1. Participants will then undergo a brain [11C]-CS1P1 PET scan
  Interventions: Drug: [11C]-CS1P1
- Participants with cognitive impairment (Alzheimer's disease): Participants with cognitive impairment will receive a single intravenous bolus injection of 12.0 - 17.0 milliCurie (mCi) of the investigational radiotracer [11C]-CS1P1. Participants will then undergo a brain [11C]-CS1P1 PET scan
  Interventions: Drug: [11C]-CS1P1

INTERVENTIONS:
Drug: [11C]-CS1P1 — Participants will receive a single intravenous bolus injection of 12.0 - 17.0 milliCurie (mCi) of the investigational radiotracer [11C]-CS1P1. Participants will then undergo a brain [11C]-CS1P1 PET scan
  Other Names: Sphingosine 1 Phosphate 1

SUMMARY:
This study involves a brain positron emission tomography (PET) scan with a new, investigational radioactive tracer called [11C]-CS1P1 to identify inflammation in the brain by testing with healthy older adults and with cognitively impaired older adults.

DETAILED DESCRIPTION:
The primary objective of this IND study is to further evaluate the [11C]-CS1P1 for PET imaging of S1P1 expression in healthy older adults and in adults with Alzheimer's disease and Related Dementia (ADRD). Investigators will complete imaging of the brain and neck in older adults with normal cognition and those with clinically diagnosed cognitive impairment from ADRD to characterize [11C]-CS1P1 uptake in the brain. Investigators will compare the normal cognition participants to patients with ADRD to collect preliminary data that will subsequently test the hypothesis that [11C]-CS1P1 uptake is elevated in patients with ADRD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any race;
* Age ≥ 50 years;
* Capable of providing written informed consent OR having a legally authorized representative (LAR) to provide informed consent for volunteering to undergo research procedure;
* Additional inclusion for ADRD group: clinical diagnosis of mild cognitive impairment or early dementia due to ADRD, OR biomarker diagnosis of Alzheimer's disease, with or without symptoms.

Exclusion Criteria:

* Hypersensitivity to [11C]-CS1P1 or any of its excipients;
* Contraindications to PET, CT, or MRI (e.g. certain incompatible electronic medical devices, inability to lie still for extended periods) that make it potentially unsafe for the individual to participate;
* Severe claustrophobia;
* Women who are currently pregnant or breast-feeding;
* Currently undergoing radiation therapy;
* Any condition that, in the opinion of the Sponsor-Investigator or designee could increase risk to the participant, limit the participant's ability to tolerate the research procedures or interfere with collection of the data (e.g., renal or liver failure, advanced cancer);
* Participants who in the last 6 months experienced any of the following cardiovascular conditions or findings in the screening electrocardiogram (ECG): clinically significant cardiac arrhythmias including high grade heart block (type 2 or greater), unstable angina, or decompensated heart failure requiring hospitalization or Class III/IV heart failure;
* Moderate to Severe anemia with Hemoglobin < than 9.9 in both males and females.
* Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.1. https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?FR=361.1

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from the community through the Volunteer for Health (VFH) Research Participant Registry at Washington University School of Medicine (WUSM), a research recruitment service offered by the Center for Clinical Studies Recruitment Enhancement Core at WUSM and through referrals from the Knight ADRC, MDC, and affiliated studies of memory and aging at Washington University, including affiliated Knight ADRC Research Imaging Program studies, referrals from physicians at Washington University and BJC Healthcare. The cohort will include healthy normal control participants and ADRD participants (n=80).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
PET imaging studies of [11C]-CS1P1 in healthy control participants and participants with Alzheimer's Disease and measuring the uptake of [11C]-CS1P1 tracer. | Through study completion, an average of 1 year
  To test the hypothesis that specific binding of [11C]-CS1P1 is elevated in participants with ADRD compared to healthy normal control participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States